CLINICAL TRIAL: NCT04458090
Title: Underutilization of Hospice in Older African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-1675; R36AG064135 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hospice Decision Making

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive hospice patient decision aid
  Interventions: Behavioral: A decision aid for patients considering Hospice care.
- Control (No Intervention): Does not receive hospice decision aid

INTERVENTIONS:
Behavioral: A decision aid for patients considering Hospice care. — A 12 page booklet and 17 min video describing hospice care
  Arms: Intervention

SUMMARY:
Despite the documented benefits of hospice, less than 2 million people utilize hospice services annually. Underuse disparities are extreme across race and ethnicity as White Americans comprise 85% of all hospice enrollees. AAs account for only 8% of hospice enrollees but are more likely to die from the top three hospice diagnoses (i.e. cancer, heart disease and dementia) than White Americans. Even when AAs enroll in hospice, they spend less time in hospice than White patients, averaging fewer than seven days in hospice care. Notably, AA hospice enrollees report a higher degree of satisfaction with end of life care when hospice is involved, as compared to AAs who are not enrolled in hospice care. There are several potential barriers that may prevent AAs from enrolling in hospice care including lack of knowledge of hospice care, mistrust in healthcare, perceived discrimination, health literacy. AAs routinely report less knowledge of hospice than White Americans, and the information that AA know about hospice often comes from non-medical professionals and is inaccurate. Some AA have persistent mistrust in healthcare due to events such as the Tuskegee Syphilis Experiments and many AA perceive discrimination when accessing healthcare. Data shows that health literacy is a stronger predictor of hospice use than race and older AAs are more likely to possess low health literacy. The driving hypothesis of this research is that by providing clear and accurate information to older AAs will help address the underutilization of hospice by clarifying misperceptions, building trust, and overcoming literacy barriers. Patient decision aids (PtDAs) are an evidence-based approach to improve patient agency in medical decision making. Research shows that AA report a desire for more agency and autonomy in decision-making yet the use of PtDAs is understudied in AA communities. This proposal offers a unique opportunity to address many of the potential barriers that may prevent older AAs from enrolling in hospice, while simultaneously expanding the literature of SDM specific to older AAs. The goals of this proposal are to evaluate if the relationships between health literacy and hospice knowledge, attitudes, and beliefs is mediated by mistrust in healthcare and perceived discrimination among AAs aged 65 or older (Aim1) and to evaluate the effect of the hospice PtDA on changing hospice knowledge and attitudes and beliefs about hospice in AA aged 65 and older (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Black or African American
* At least 65 years of age

Exclusion Criteria:

* Non-English speakers.
* Patients with cognitive Impairments preventing ability to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channing E Tate, MPH, PhD(c), Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tate CE, Perez-Jolles M, Scherer LD, Shiferaw T, Mami G, Matlock DD, Huebschmann AG. "Hospice was Created by the KKK"-Black Americans' Perspectives on Hospice Care. J Racial Ethn Health Disparities. 2025 Feb 27. doi: 10.1007/s40615-025-02340-w. Online ahead of print. PMID 40014286
- [Derived] Brereton E, Harger G, Matlock DD, Dorsey Holliman B, Tate CE. How Do Patients Describe Hospice Care? A Qualitative Analysis of the Language Used by Older Adults to Describe Hospice Care. J Palliat Med. 2022 Nov;25(11):1692-1696. doi: 10.1089/jpm.2022.0011. Epub 2022 Aug 9. PMID 35944273
- [Derived] Tate CE, Venechuk G, Pierce K, Khazanie P, Ingle MP, Morris MA, Allen LA, Matlock DD. Development of a Decision Aid for Patients and Families Considering Hospice. J Palliat Med. 2021 Apr;24(4):505-513. doi: 10.1089/jpm.2020.0250. Epub 2021 Jan 13. PMID 33439075

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 72 | 72
Completed | 72 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 72 | 72 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 72 | 144
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 72 | 144
Hospice Knowledge Test [Mean (Full Range); unit: units on a scale] — Hospice Knowledge Scale is a 23-item true/false scale. Each question is worth 1 point with 23 being the highest score. Higher scores indicate more hospice knowledge. Absolute scores were measured at baseline and 1 month follow-up.
  units on a scale | 17 [0 to 23] | 17 [0 to 23] | 17 [0 to 23]
Hospice Beliefs and Attitudes Scale [Mean (Full Range); unit: units on a scale] — Hospice Attitudes and Beliefs Scale is an 8-item 5-point Likert scale (ranging from Strongly Agree to Strongly Disagree). Each question is scored based on 5 point scale. Maximum score 40 and minimum score 8. Higher scores indicate more favorable opinions of hospice. Absolute scores were measured at baseline and 1 month follow-up.
  units on a scale | 28 [11 to 38] | 27 [12 to 40] | 27.5 [11 to 40]
Decision Self-Efficacy Scale [Mean (Full Range); unit: units on a scale] — Decision Self-Efficacy Scale is an 11-item 5-point Likert scale (ranging from not at all confident to very confident). Maximum score is 100 and minimum score is 0. Higher scores indicate more self-efficacy. Absolute scores were measured at baseline and 1 month follow-up.
  units on a scale | 78 [0 to 100] | 72 [0 to 100] | 75 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Hospice Knowledge Scale
Description: Hospice Knowledge Scale is a 23-item true/false scale. Each question is worth 1 point with 23 being the highest score. Possible scores range from 0 to 23, with higher scores indicate more hospice knowledge.
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 72
units on a scale | 17 [0 to 23] | 17 [0 to 23]

2. Primary Outcome: Hospice Attitudes and Beliefs Scale
Description: Hospice Attitudes and Beliefs Scale is an 8-item 5-point Likert scale (ranging from Strongly Agree to Strongly Disagree). Each question is scored based on 5 point scale. Maximum score 40 and minimum score 8. Higher scores indicate more favorable opinions of hospice.
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 72
units on a scale | 31 [9 to 40] | 30 [9 to 40]

3. Primary Outcome: Decision Self Efficacy Scale
Description: Decision Self-Efficacy Scale is an 11-item 5-point Likert scale (ranging from not at all confident to very confident). Maximum score is 100 and minimum score is 0. Higher scores indicate more self-efficacy.
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 72
units on a scale | 89 [48 to 100] | 78 [11 to 100]

ADVERSE EVENTS:
Description: Minimal risk study only collecting survey date and All Cause Mortality, Serious Adverse Events, and other adverse events were not monitored.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT04458090/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04458090/ICF_001.pdf